CLINICAL TRIAL: NCT05369663
Title: Effects of Personal Protective Equipment on Speech Acoustics
Brief Title: Personal Protective Equipment Effects
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, ahmet mutlu, asistant professor, Istanbul Medeniyet University
Other Study IDs: Effects on speech acoustics
Record Dates: First submitted 2022-04-25; First posted 2022-05-11 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Speech Disorders; Voice Disorders
Keywords: speech acoustics
MeSH Terms: conditions — Speech Disorders; Voice Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- no mask: no mask use
- surgical mask: surgical mask use
  Interventions: Device: mask use
- N99 mask: N99 mask use
  Interventions: Device: mask use
- face shield: face shield use
  Interventions: Device: mask use
- surgical mask+ faceshield: surgical mask+ faceshield use
  Interventions: Device: mask use
- N99 mask+ faceshield: N99 mask+ faceshield use
  Interventions: Device: mask use

INTERVENTIONS:
Device: mask use — face mask use
  Groups: N99 mask; N99 mask+ faceshield; face shield; surgical mask; surgical mask+ faceshield

SUMMARY:
Severe acute respiratory syndrome coronavirus-2 transmits through droplets; thus, oral, nasal, and conjunctival mucosas are related to contamination, and wearing personal protective equipment (PPE) is strongly suggested. Several communication problems between the patient and healthcare workers related to PPE use are reported. In this study, investigators aimed to investigate changes in the acoustic parameters of speech sounds when different PPE are used.

DETAILED DESCRIPTION:
It was planned as a cross-sectional study enrolled 18 healthy male and female participants. After the informed consent, participants were asked to pronounce a [ɑː] vowel for at least 3 seconds for voice quality estimation. Afterward, all Turkish vowels were produced for a minimum of 200 ms. Finally, three Turkish fricative consonants ([f], [s], [ʃ]) were produced in consonant/vowel/consonant format and in different vowel contexts within a carrier sentence. Recordings were repeated for the following conditions: no PPE, surgical-mask, N99-mask, face shield, surgical-mask+faceshield, and N99+faceshield. All recordings were analyzed with proper statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* native Turkish speakers

Exclusion Criteria:

* having an acute respiratory system infection history of any vocal fold surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals. Based on health caregiving people (doctors, nurses)
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-01-16 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
The change on voice acoustics due to different personal protective equipments use | 1 months
  speech material for six different conditions: no PPE,surgical mask,N99 mask,face shield,surgical mask+ face shield, N99+face shield were recorded with a microphone.Recordings were performed in a random order. Obtained speech records were segmented according to the speech material and saved. Each of the segmented files was analyzed using Praat software and related scripts. The voice quality parameters were estimated on sustained [ɑː] vowels via Praat software (Praat is an open source software which enables voice acoustics analysis). Mean values of the different formant frequencies and formant bandwidth frequency values at midpoints of the analyzed segments of the vowels were measured. Spectral moments of the consonants were measured. The formant and spectral moment were measured using Praat scripts. All outcome measurements are in Hertz (Hz), so all measurements are held in primary outcome 1 measure section.

CONTACTS AND LOCATIONS:
Overall Officials: ahmet mutlu, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gama R, Castro ME, van Lith-Bijl JT, Desuter G. Does the wearing of masks change voice and speech parameters? Eur Arch Otorhinolaryngol. 2022 Apr;279(4):1701-1708. doi: 10.1007/s00405-021-07086-9. Epub 2021 Sep 22. PMID 34550454